CLINICAL TRIAL: NCT02919917
Title: Treatment of Post-SCI Hypotension: A Randomized Controlled Study of Usual Care Versus Anti Hypotension Therapy
Brief Title: Treatment of Post-SCI Hypotension
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Jill M. Wecht, Ed.D., Principal Invesitgator, James J. Peters Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WEC-16-050
Record Dates: First submitted 2016-09-22; First posted 2016-09-30 (Estimated); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Spinal Cord Injury; Autonomic Dysreflexia; Orthostatic Hypotension; Baroreceptor Integrity; Sympathetic Integrity; Vagal Integrity; Hypotension; Cerebral Blood Flow; Blood Pressure; Venous Occlusion Plethysmography
MeSH Terms: conditions — Spinal Cord Injuries; Autonomic Dysreflexia; Hypotension, Orthostatic; Hypotension | interventions — Midodrine

STUDY DESIGN:
Intervention Model Description: Newly injured individuals with SCI will be eligible to participate if they demonstrate hypotension (systolic blood pressure </= 110 mmHg in males or </= 100 mmHg in females) upon admission to acute in-patient rehabilitation at Mount Sinai Medical Center, New York, NY. Eligible participants will be randomized to usual care (administered anti-hypotensive therapy only if they demonstrate symptoms of hypotension: dizziness, lightheadedness, nausea, blurred vision, syncope) or treatment of hypotension based on a systolic blood pressure below the hypotensive threshold. Time spent in active rehabilitation program will be compared between the usual care and treatment groups.
Who Masked: Care Provider
Masking Description: Therapists administering rehabilitation will be blinded to the randomization of patients enrolled in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care Group (Experimental): Individuals randomized to the usual care group will receive BP management according to the usual care in current practice in the SCI Rehabilitation Unit.
  Will receive treatment only if they experience symptoms that are associated with low BP (dizziness, lightheadedness, nausea, blurry vision, loss of consciousness, etc.).
  Treatment to lessen or eliminate these symptoms of low blood pressure will be guided by the attending physician and can include physical countermeasures to increase blood pressure (abdominal binders, comperssion stockings, etc.) and/or midodrine .
  Interventions: Drug: Midodrine Hydrochloride
- BP Threshold Treatment Group (Experimental): Individuals assigned to the BP threshold treatment group will receive BP management, regardless of symptoms, to maintain systolic BP between 111-135 mmHg for males and 101-135 mmHg for females for the duration of their in-patient hospital stay.
  This treatment will be started based on your low BP, regardless of if you experience symptoms that are associated with low BP (dizziness, lightheadedness, nausea, blurry vision, loss of consciousness, etc.). Before you start on any medication you will receive physical countermeasures to increase blood pressure (abdominal binders, comperssion stockings, etc.).
  If your blood pressure remains low after using these countermeasures you will begin to take midodrine 3 times a day as described in the intervention section. The dosage will increase and be stopped once until your seated SBP is between 111-135 mmHg.
  Interventions: Drug: Midodrine Hydrochloride

INTERVENTIONS:
Drug: Midodrine Hydrochloride — Level 1: Compression stockings, abdominal binder Level 2: Midodrine 5mg 2x/d Level 3: Midodrine 10mg 2x/d Level 4: Midodrine 15mg 2x/d Level 5: Midodrine 20mg 2x/d Level 6 Midodrine 20mg 2x/d and Fludrocortisone 0.1mg 2x/d Level 7 Midodrine 20mg 2x/d and Fludrocortisone 0.2mg 2x/d
  Other Names: Midodrine
  Arms: BP Threshold Treatment Group
Drug: Midodrine Hydrochloride — Level 1: Compression stockings, abdominal binder Level 2: Midodrine 5mg 2x/d Level 3: Midodrine 10mg 2x/d Level 4: Midodrine 15mg 2x/d Level 5: Midodrine 20mg 2x/d Level 6 Midodrine 20mg 2x/d and Fludrocortisone 0.1mg 2x/d Level 7 Midodrine 20mg 2x/d and Fludrocortisone 0.2mg 2x/d
  Other Names: Midodrine
  Arms: Usual Care Group

SUMMARY:
While treatment strategies for OH have been identified for use in persons with acute SCI, the field of SCI medicine lacks a gold standard for treatment thresholds and well-defined outcome parameters. Comprehensively documenting the impact of orthostatic hypotension (OH), regardless of symptoms, during acute rehabilitation and identifying the effects of two different treatment approaches on therapy participation and adherence to an intended rehabilitation plan could have a significant impact on clinical practice in the acute rehabilitation setting following SCI.

DETAILED DESCRIPTION:
Baseline Testing: Subjects will visit the testing laboratory on the SCI Rehabilitation Unit for baseline data collection, prior to initiation of the treatment protocol. Upon arrival, subjects will be placed in the supine position on an adjustable surface for instrumentation, which will be conducted in a quiet, dimly lit, thermo-neutral testing environment. After a 20-minute period of quiet rest, a 10-minute sample of supine heart rate (HR), respiratory rate, BP and CBF velocity data will be collected. Venous occlusion plethysmography (Vop) will be collected in the supine position for two 5-minute periods. After the supine data collection, subjects will be passively moved into the seated position, with the knees and hips at 90°, for the 10-minute seated data collection period. Subjects will be asked to complete two surveys related to AD and OH symptomology. Finally, subjects will be fitted with a 24-hour HR and BP monitor and will be asked to go about their normal routine. A record of all daily activities including rehabilitation, medications, eating and sleep/wake times will be logged. This testing session should take approximately 1 hour.

Daily Testing: Every day supine and seated BP measurements will be performed at least three times per day. These BP assessments will be recorded in the supine and seated positions in the subject's room by a patient care associate who is blind to the study arm allocation. For every scheduled physical and occupational therapy session, the treating therapist will be asked to complete a brief 6 question survey to document if that session was altered, disrupted, or missed due to hypotension (Therapist Reported Version). The subject will also be asked to complete a brief survey to determine if from their perspective the session was altered, disrupted or missed due to hypotension (Subject Reported Version). In addition, every day a co-investigator and the attending physician for that subject will complete an EMR review of queried BP values within the previous 24 hours, symptoms of low BP, adverse events related to high or low BP, and will review (and act upon for the usual care arm) the protocol treatment decision tree.

Weekly Testing: At weekly intervals of between 6 and 8 days, subjects will be asked to visit the testing laboratory on the SCI Rehabilitation Unit. Procedures for the weekly testing sessions will be the same as for the Baseline Testing. The 24-hour BP assessment will be conducted twice weekly.

Discharge Testing: At discharge subjects will undergo similar testing as described during the Baseline and Weekly Testing with the addition of the Patient Global Impression of Change survey, which will be administered by the Mount Sinai Site Research Assistant.

ELIGIBILITY:
Inclusion Criteria:

* Any level of injury;
* Any AIS grade of SCI;
* Non-ventilator dependent
* Primarily wheelchair dependent for mobility;
* Duration of injury < 1 year
* Systolic BP less than 110 mmHg and/or diastolic BP less than 70 mmHg for males.
* Systolic BP less than 100 mmHg and/or diastolic BP less than 70 mmHg for females
* Primary Language is English.
* Able to provide informed consent

Exclusion Criteria:

* Have insufficient mental capacity to independently provide informed consent
* Have insufficient English speaking or reading ability to provide informed consent or complete assessments in English
* Have contraindications to the use of midodrine hydrochloride
* Are pregnant

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill M Wecht, Ed.D., Principal Investigator — James J. Peters VA Medical Center
Locations (2):
- United States (2):
  - Mount Sinai School of Medicine, New York, New York
  - VA Medical Center, Bronx, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Wecht JM, Weir JP, Huang V, Escalon MX, Bryce TN. Treatment of Orthostatic Hypotension During Acute Inpatient Rehabilitation After Spinal Cord Injury: Usual Care vs. Anti-hypotensive Therapy. Am J Hypertens. 2024 Jul 15;37(8):554-560. doi: 10.1093/ajh/hpae057. PMID 38712567
- [Derived] Vaccaro DH, Weir JP, Noonavath M, Bryce TN, Escalon MX, Huang V, Delgado A, Wecht JM. Orthostatic systemic and cerebral hemodynamics in newly injured patients with spinal cord injury. Auton Neurosci. 2022 Jul;240:102973. doi: 10.1016/j.autneu.2022.102973. Epub 2022 Mar 18. PMID 35366432

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care Group: Individuals randomized to the usual care group will receive BP management according to the usual care in current practice in the SCI Rehabilitation Unit.
  Will receive treatment only if they experience symptoms that are associated with low BP (dizziness, lightheadedness, nausea, blurry vision, loss of consciousness, etc.).
  Treatment to lessen or eliminate these symptoms of low blood pressure will be guided by the attending physician and can include physical countermeasures to increase blood pressure (abdominal binders, comperssion stockings, etc.) and/or midodrine .
  Midodrine Hydrochloride: Level 1: Compression stockings, abdominal binder Level 2: Midodrine 5mg 2x/d Level 3: Midodrine 10mg 2x/d Level 4: Midodrine 15mg 2x/d Level 5: Midodrine 20mg 2x/d Level 6 Midodrine 20mg 2x/d and Fludrocortisone 0.1mg 2x/d Level 7 Midodrine 20mg 2x/d and Fludrocortisone 0.2mg 2x/d
- BP Threshold Treatment Group: Individuals assigned to the BP threshold treatment group will receive BP management, regardless of symptoms, to maintain systolic BP between 111-135 mmHg for males and 101-135 mmHg for females for the duration of their in-patient hospital stay.
  This treatment will be started based on your low BP, regardless of if you experience symptoms that are associated with low BP (dizziness, lightheadedness, nausea, blurry vision, loss of consciousness, etc.). Before you start on any medication you will receive physical countermeasures to increase blood pressure (abdominal binders, comperssion stockings, etc.).
  If your blood pressure remains low after using these countermeasures you will begin to take midodrine 3 times a day as described in the intervention section. The dosage will increase and be stopped once until your seated SBP is between 111-135 mmHg.
  Midodrine Hydrochloride: Level 1: Compression stockings, abdominal binder Level 2: Midodrine 5mg 2x/d Level 3: Midodrine 10mg 2x/d Level 4: Midodrine 15mg 2x/d Level 5: Midodrine 20mg 2x/d Level 6 Midodrine 20mg 2x/d and Fludrocortisone 0.1mg 2x/d Level 7 Midodrine 20mg 2x/d and Fludrocortisone 0.2mg 2x/d
Period: Overall Study
Arm/Group | Usual Care Group | BP Threshold Treatment Group
Started | 33 | 33
Completed | 29 | 25
Not Completed | 4 | 8
Not completed — Withdrawal by Subject | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care Group | BP Threshold Treatment Group | Total
Number analyzed (Participants) | 29 | 25 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 23 | 21 | 44
  >=65 years | 6 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.82 (17.49) | 41.97 (15.84) | 43.89 (16.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 24 | 19 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 7 | 15
  White | 10 | 10 | 20
  More than one race | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 25 | 54

OUTCOME MEASURES:

1. Primary Outcome: Affected Therapy Sessions
Description: Responses to the questions "was the therapy session affected by low BP or concern for low BP development?" between the usual care and BP threshold treatment groups. The percent of sessions with a "yes" response are reported.
Time Frame: Inpatient hospitalization (up to 4 months)
Measure: Number; unit: percentage of sessions
Units Other Than Participants: Number of therapy sessions
Arm/Group | Usual Care Group | BP Threshold Treatment Group
Number analyzed (Participants) | 29 | 25
Number analyzed (Number of therapy sessions) | 1123 | 1258
percentage of sessions | 16.4 | 10.9

2. Primary Outcome: Systolic Blood Pressure
Description: Systolic hypertension (>/= 140 mmHg)
Time Frame: Inpatient hospitalization (up to 4 months)
Measure: Number; unit: percentage of BP assessments
Units Other Than Participants: total BP assessments
Arm/Group | Usual Care Group | BP Threshold Treatment Group
Number analyzed (Participants) | 33 | 33
Number analyzed (total BP assessments) | 1574 | 1940
percentage of BP assessments | 4.8 | 5.3

3. Secondary Outcome: Systolic Blood Pressure
Description: Systolic hypotension (males: < 110 mmHg; females: < 100 mmHg)
Time Frame: Inpatient Hospitalizations (up to 4 months)
Measure: Number; unit: percentage of BP assessments
Units Other Than Participants: Total BP assessments
Arm/Group | Usual Care Group | BP Threshold Treatment Group
Number analyzed (Participants) | 33 | 33
Number analyzed (Total BP assessments) | 1574 | 1940
percentage of BP assessments | 39.7 | 43.0

4. Secondary Outcome: Missed Therapy Sessions
Description: Percentages of missed therapy sessions, due to low BP or concern for low BP development, in the usual care and BP treatment groups
Time Frame: Inpatient Hospitalizations (up to 4 months)
Measure: Number; unit: percentage of missed therapy sessions
Units Other Than Participants: Number of interrupted sessions
Arm/Group | Usual Care Group | BP Threshold Treatment Group
Number analyzed (Participants) | 29 | 25
Number analyzed (Number of interrupted sessions) | 314 | 212
percentage of missed therapy sessions | 58.60 | 65.8

ADVERSE EVENTS:
Time Frame: Inpatient Hospitalizations (up to 4 months)
Description: No higher risk of SAE or all-cause mortality in the usual care or BP treatment groups compared to expected for this population.
Arm/Group | Usual Care Group | BP Threshold Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/25
Other Adverse Events (participants affected / at risk) | 0/29 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/17/NCT02919917/Prot_SAP_ICF_000.pdf